CLINICAL TRIAL: NCT02341664
Title: Patient and Provider Assessment of Lipid Management Registry
Acronym: PALM
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00058405
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Hyperlipidemia; Hypercholesterolemia; Cardiovascular Disease; Diabetes; Chronic Kidney Disease (CKD); Hypertension; Smoking; Myocardial Infarction (MI); Unstable Angina; Angina; Coronary Artery Disease (CAD); Stroke; Transient Ischemic Attack (TIA); Carotid Stenosis; Peripheral Arterial Disease; Atherosclerosis; Claudication
Keywords: Mobile Tablet Device; Outpatient Clinic; Tobacco; Health; Barriers; Prevention; Prescribing Practices; Informed Consent; Statin; Lipid Panel; Low Density Lipoprotein-C; Blood Draw; ACC/AHA Guidelines; Adult Treatment Panel Guidelines (ATPIII); Atherosclerotic Cardiovascular Disease (ASCVD); Cholesterol-lowering therapies; Cholesterol Management; Cardiovascular Risk; 10-year CVD Risk; Labs; Coronary revascularization; Arterial revascularization; Imaging
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia; Cardiovascular Diseases; Diabetes Mellitus; Renal Insufficiency, Chronic; Hypertension; Smoking; Myocardial Infarction; Angina, Unstable; Angina Pectoris; Coronary Artery Disease; Stroke; Ischemic Attack, Transient; Carotid Stenosis; Peripheral Arterial Disease; Atherosclerosis; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the Patient and Provider Assessment of Lipid Management Registry (PALM) is to gain a better understanding of physicians' cholesterol medication prescribing practices, patient and physician attitudes and beliefs related to cholesterol management, and current utilization of cholesterol-lowering therapies given the new ACC/AHA guideline recommendations. The PALM Registry hopes to allow for the design of ways to improve cholesterol management and decrease the burden of cardiovascular disease (CVD) in the US.

DETAILED DESCRIPTION:
The PALM registry is a multicenter, observational registry aimed at evaluating how cholesterol management is applied in current clinical practice. This registry will recruit approximately 175 sites in the United States to enroll 7,500 patients with cardiovascular risk factors warranting consideration of lipid-lowering therapies as well as those already on statin therapy. Enrolling clinicians will include primary care providers, internal medicine providers, family medicine providers, cardiologists, and endocrinologists. Site selection will also target geographic diversity to ensure representation from all regions of the U.S., including rural and urban areas, as well as from minority populations. This registry is unique featuring the use of a mobile tablet-based enrollment device. This tablet-based enrollment tool is designed to adapt to the workflow of an outpatient practice, allowing research procedures (including screening, informed consent and patient survey) to be carried out during the patient visit, and maximizes paper-less data entry. All patient management decisions (including the choice of cholesterol-lowering therapy) are completely at the discretion of the care providers. This registry will involve retrospective and prospective patient data collection. Baseline data from patients and physicians will be collected. There will be no patient follow-up.

The target sample size (n=7,500) in this registry is not determined based on statistical considerations, but is based upon a non-probabilistic sampling approach, in order to obtain sufficient exposure data in patients who are in the various atherosclerotic cardiovascular disease (ASCVD) risk groups. During the enrollment period, balance across groups will be maintained by frequent monitoring of enrollment. Adaptive enrollment and capping will be considered to ensure adequate exposure across groups, physician type, and geographic location. Data quality will be assured by web-based or application-based data collection tool queries and data quality reports . Data quality control measures will include: data entry missing and range checks, data validation checks; standard record level checks that are run on the database to identify suspected duplicate, blank, or missing records; and logic checks and data surveillance of trends in data entry and query processing. The tools will prompt user to correct any missing, out of range, or potentially incorrect data. There are no interventions, no outside monitoring of sites nor a DSMB with this registry.

ELIGIBILITY:
Inclusion Criteria:

1. Prior evidence of clinical atherosclerotic cardiovascular disease (ASCVD) which can include any of the following:

   * Hospitalization for acute myocardial infarction or unstable angina
   * Coronary revascularization or chronic coronary artery disease with or without angina
   * Other arterial (carotid, abdominal, renal or lower extremity) revascularization (e.g., surgical bypass, percutaneous intervention, arterial vascular reconstruction, abdominal aortic aneurysm repair, excluding dialysis fistulas or arteriovenous grafts).
   * Ischemic stroke or transient ischemic attack (TIA)
   * Imaging evidence of > 70% diameter stenosis in any carotid artery or clinical documentation of severe carotid stenosis
   * Peripheral arterial disease secondary to atherosclerosis (e.g., aortic aneurysm, ankle brachial index <0.9, imaging evidence of >50% diameter stenosis in any peripheral artery, or claudication)
2. Currently on statin therapy
3. Low density lipoprotein cholesterol (LDL-C) level ≥ 130 mg/dL within the last 2 years (treated or untreated)
4. Age ≥ 65 years
5. Age ≥ 40 years with at least 1 of the following:

   * Diabetes
   * Chronic Kidney Disease (CKD), defined as eGFR <60 ml/min or documented stage III or higher CKD
   * 10-year ASCVD risk ≥ 5% (per the 2013 ACC/AHA Guideline on the Assessment of Cardiovascular Risk)
   * 2 or more of the following characteristics: Male sex; Systolic BP > 140 mmHg or on medication for hypertension; Current tobacco use

Exclusion Criteria:

1. Unable or unwilling to provide informed consent, including but not limited to cognitive or language barriers (reading or comprehension)
2. Anticipated life expectancy less than 6 months
3. Participation in any clinical trial involving a medical treatment at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry will recruit approximately 175 sites to enroll ~7,500 patients with cardiovascular risk factors warranting consideration of lipid-lowering therapies as well as those already on statin therapy. Patients will be recruited from outpatient clinics including primary care, internal medicine, family medicine, cardiology, and endocrinology. Patients will be recruited across all regions of the U.S., including rural and urban areas, as well as from minority populations.
Sampling Method: Non-Probability Sample
Enrollment: 7658 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Lipid-lowering therapy use among a contemporary, nationally representative, community-based sample of adult patients receiving primary and subspecialty care in the US. | baseline, upon enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Wang, MD, Principal Investigator — Duke Clinical Research Institute; Eric Peterson, MD, Principal Investigator — Duke Clinical Research Institute
Locations (14):
- United States (14):
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - COR Healthcare, San Pedro, California
  - Ventura Cardiology Consultants Medical Group, Inc, Ventura, California
  - Maya Research Center, Inc, Hialeah, Florida
  - Wellness Clinical Research, LLC, Hialeah Gardens, Florida
  - Infinity Clinical Research, Plantation, Florida
  - Midwest Heart and Vascular Specialists, LLC, Overland Park, Kansas
  - Krishnan Challappa, MD, PSC, Elizabethtown, Kentucky
  - HealthEast Clinical Trials Office, Saint Paul, Minnesota
  - Long Island Heart Associates, Mineola, New York
  - Gotham Cardiovascular Research, New York, New York
  - New Bern Internal Medicine, New Bern, North Carolina
  - Detweiler Family Medicine Associates, PC, Lansdale, Pennsylvania
  - Charleston Internal Medicine, Inc., Charleston, West Virginia

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: prevalence, treatment, and control of high levels of low-density lipoprotein cholesterol--United States, 1999-2002 and 2005-200. MMWR Morb Mortal Wkly Rep. 2011 Feb 4;60(4):109-14. PMID 21293326
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] Goff DC Jr, Lloyd-Jones DM, Bennett G, Coady S, D'Agostino RB, Gibbons R, Greenland P, Lackland DT, Levy D, O'Donnell CJ, Robinson JG, Schwartz JS, Shero ST, Smith SC Jr, Sorlie P, Stone NJ, Wilson PW, Jordan HS, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the assessment of cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S49-73. doi: 10.1161/01.cir.0000437741.48606.98. Epub 2013 Nov 12. No abstract available. PMID 24222018
- [Background] Wanner C, Tonelli M; Kidney Disease: Improving Global Outcomes Lipid Guideline Development Work Group Members. KDIGO Clinical Practice Guideline for Lipid Management in CKD: summary of recommendation statements and clinical approach to the patient. Kidney Int. 2014 Jun;85(6):1303-9. doi: 10.1038/ki.2014.31. Epub 2014 Feb 19. PMID 24552851
- [Background] Jellinger PS, Smith DA, Mehta AE, Ganda O, Handelsman Y, Rodbard HW, Shepherd MD, Seibel JA; AACE Task Force for Management of Dyslipidemia and Prevention of Atherosclerosis. American Association of Clinical Endocrinologists' Guidelines for Management of Dyslipidemia and Prevention of Atherosclerosis. Endocr Pract. 2012 Mar-Apr;18 Suppl 1:1-78. doi: 10.4158/ep.18.s1.1. No abstract available. PMID 22522068
- [Background] Pencina MJ, Navar-Boggan AM, D'Agostino RB Sr, Williams K, Neely B, Sniderman AD, Peterson ED. Application of new cholesterol guidelines to a population-based sample. N Engl J Med. 2014 Apr 10;370(15):1422-31. doi: 10.1056/NEJMoa1315665. Epub 2014 Mar 19. PMID 24645848
- [Background] Lab's HIE solution connects LIS to EMR and HIS. MLO Med Lab Obs. 2009 Dec;41(12):30, 32-4. No abstract available. PMID 20085087
- [Background] Mosca L, Linfante AH, Benjamin EJ, Berra K, Hayes SN, Walsh BW, Fabunmi RP, Kwan J, Mills T, Simpson SL. National study of physician awareness and adherence to cardiovascular disease prevention guidelines. Circulation. 2005 Feb 1;111(4):499-510. doi: 10.1161/01.CIR.0000154568.43333.82. PMID 15687140
- [Background] Wei MY, Ito MK, Cohen JD, Brinton EA, Jacobson TA. Predictors of statin adherence, switching, and discontinuation in the USAGE survey: understanding the use of statins in America and gaps in patient education. J Clin Lipidol. 2013 Sep-Oct;7(5):472-83. doi: 10.1016/j.jacl.2013.03.001. Epub 2013 Mar 13. PMID 24079289
- [Background] Desai CS, Martin SS, Blumenthal RS. Non-cardiovascular effects associated with statins. BMJ. 2014 Jul 17;349:g3743. doi: 10.1136/bmj.g3743. PMID 25035309
- [Background] Zhang H, Plutzky J, Skentzos S, Morrison F, Mar P, Shubina M, Turchin A. Discontinuation of statins in routine care settings: a cohort study. Ann Intern Med. 2013 Apr 2;158(7):526-34. doi: 10.7326/0003-4819-158-7-201304020-00004. PMID 23546564
- [Background] Gagne JJ, Choudhry NK, Kesselheim AS, Polinski JM, Hutchins D, Matlin OS, Brennan TA, Avorn J, Shrank WH. Comparative effectiveness of generic and brand-name statins on patient outcomes: a cohort study. Ann Intern Med. 2014 Sep 16;161(6):400-7. doi: 10.7326/M13-2942. PMID 25222387
- [Derived] Fanaroff AC, Li S, Webb LE, Miller V, Navar AM, Peterson ED, Wang TY. An Observational Study of the Association of Video- Versus Text-Based Informed Consent With Multicenter Trial Enrollment: Lessons From the PALM Study (Patient and Provider Assessment of Lipid Management). Circ Cardiovasc Qual Outcomes. 2018 Apr;11(4):e004675. doi: 10.1161/CIRCOUTCOMES.118.004675. PMID 29625993
- [Derived] Navar AM, Wang TY, Goldberg AC, Robinson JG, Roger VL, Wilson PF, Virani SS, Elassal J, Lee LV, Webb LE, Peterson E. Design and rationale for the Patient and Provider Assessment of Lipid Management (PALM) registry. Am Heart J. 2015 Nov;170(5):865-71. doi: 10.1016/j.ahj.2015.08.002. Epub 2015 Aug 7. PMID 26542493